CLINICAL TRIAL: NCT00939276
Title: Macular Edema Incidence/Severity Reduction With Nevanac
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient recruitment difficulties
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-003; EudraCT Number: 2009-010536-17
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Diabetic Retinopathy
Keywords: cataract surgery; macular edema; prevention
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEVANAC (Experimental): One drop instilled in the study eye 3 times daily (morning, midafternoon, and bedtime) beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery
  Interventions: Drug: Nepafenac ophthalmic suspension, 0.1% (NEVANAC®)
- Nepafenac Vehicle (Placebo Comparator): One drop instilled in the study eye 3 times daily (morning, midafternoon, and bedtime) beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery
  Interventions: Drug: Nepafenac ophthalmic suspension vehicle

INTERVENTIONS:
Drug: Nepafenac ophthalmic suspension, 0.1% (NEVANAC®) — One drop instilled in the study eye 3 times daily (morning, midafternoon, and bedtime) beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery
  Other Names: NEVANAC®
  Arms: NEVANAC
Drug: Nepafenac ophthalmic suspension vehicle — One drop instilled in the study eye 3 times daily (morning, midafternoon, and bedtime) beginning the day before surgery, continuing on the day of surgery and through the first 90 days following surgery
  Arms: Nepafenac Vehicle

SUMMARY:
The purpose of this study is to evaluate NEVANAC in patients with diabetic retinopathy who developed macular edema (ME) within 90 days following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens (IOL) into the lens capsule.
* History of Type 1 or Type 2 diabetes.
* History of nonproliferative diabetic retinopathy (NPDR), mild, moderate, or severe, in the study eye as defined by the International Clinical Diabetic Retinopathy Disease Severity Scale.
* Able to understand and sign an informed consent approved by an IRB/IEC.
* Central subfield macular thickness less than or equal to 320 μm in the study eye prior to cataract surgery.
* Absence of clinically significant macular edema in the study eye as detected by clinical exam.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Signs of vitreomacular traction or epiretinal membrane in the study eye as detected by the reading center or Investigator.
* Current or previous ocular disease other than diabetic retinopathy in the study eye that, in the opinion of the Investigator, would have confounded the assessments of the macula, the retina, or central vision.
* Planned multiple procedures for the study eye during the cataract/IOL implantation surgery (eg, trabeculoplasty, corneal transplant).
* Corneal transplant in study eye.
* Baseline cumulative corneal fluorescein staining score (ie, sum of scores for all 5 corneal regions) for the study eye greater than or equal to 5, or baseline corneal fluorescein staining score in any single region for the study eye greater than or equal to 3.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who develop macular edema within 90 days following cataract surgery | Time to event

SECONDARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) from baseline to Day 90 | Baseline, Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Pollack A, Staurenghi G, Sager D, Mukesh B, Reiser H, Singh RP. Prospective randomised clinical trial to evaluate the safety and efficacy of nepafenac 0.1% treatment for the prevention of macular oedema associated with cataract surgery in patients with diabetic retinopathy. Br J Ophthalmol. 2017 Apr;101(4):423-427. doi: 10.1136/bjophthalmol-2016-308617. Epub 2016 Jul 7. PMID 27388251